CLINICAL TRIAL: NCT07110688
Title: Novel Multimodal Neural, Physiological, and Behavioral Sensing and Machine Learning for Mental States
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Maryam Shanechi, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R61MH135407 (NIH); R61MH135407 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-08-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: No Condition; Study Mental State in Healthy Populations and Drug-resistant Epilepsy Patients With Existing iEEG
Keywords: neurotechnology; neuropsychiatric disorders; brain-machine interface

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral tasks to assess mental states (Experimental)
  Interventions: Behavioral: Virtual human social interaction; Behavioral: Cold pressor test

INTERVENTIONS:
Behavioral: Virtual human social interaction — The participants will perform a social interaction with the virtual human agent platform to assess mental states.
Behavioral: Cold pressor test — Healthy participants will immerse one hand in cold water for less than 3 minutes, while physiological data will be collected by the new wearable sensor from the other hand.

SUMMARY:
In this program, the investigators will develop novel multimodal neural-behavioral-physiological monitoring tools (software and hardware), and machine learning models for mental states within social processes and beyond. The tools consist of a multimodal skin-like wearable sensor for physiological and biochemical sensing; a conversational virtual human platform to evoke naturalistic social processes; audiovisual affect recognition software; synchronization tools; and machine learning methods to model the multimodal data. The investigators will demonstrate the tools in healthy subjects without neural recordings and in patients with drug-resistant epilepsy who already have intracranial EEG (iEEG) electrodes implanted based on clinical criteria for standard monitoring to localize seizures, which is unrelated to our study.

ELIGIBILITY:
For the healthy population, all subjects over the age of 18 who are able and willing to give informed consent will be eligible.

For the epilepsy population, inclusion criteria are:

* Patients who suffer from drug-resistant epilepsy and already have intracranial EEG (iEEG) electrodes implanted based on clinical criteria for their standard seizure localization (unrelated to our study) will be eligible. Most patients are healthy adults outside of their epilepsy.
* Subjects >= 18 are only included in this study.
* All patients with the above conditions and with already-implanted electrodes who are willing to participate and able to cooperate and follow research instructions will be recruited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | 7-10 days
  Momentary self-reports of the Positive and Negative Affect Schedule (PANAS) will be administered in a tablet-based application, which measures momentary positive and negative affect. These self-reports return scores indicative of momentary mental state. Self-reports are obtained intermittently from the participants.
Visual Analog Scale (VAS) | 7-10 days
  Momentary self-reports of the Visual Analog Scale (VAS) of depression, anxiety, and energy will be administered in a tablet-based application. These are fast self-reports to indicate the affect level along a line from none to prominent. These self-reports return scores indicative of momentary mental state. Self-reports are obtained intermittently from the participants.
Hamilton Depression Rating Scales (HAMD-6) | 7-10 days
  Momentary self-reports of Hamilton Depression Rating Scales (HAMD-6) will be administered in a tablet-based application, which is widely used to measure the severity of the depressive state. These self-reports return scores indicative of momentary mental state. Self-reports are obtained intermittently from the participants.
Hamilton Anxiety Rating Scales (HAM-A) | 7-10 days
  Momentary self-reports of Hamilton Anxiety Rating scales (HAM-A) will be administered in a tablet-based application, which is widely used to measure the severity of the anxiety state. These self-reports return scores indicative of momentary mental state. Self-reports are obtained intermittently from the participants.
Immediate Mood Scalar (IMS) | 7-10 days
  Momentary self-reports of the Immediate Mood Scalar (IMS) will be administered in a tablet-based application, which measures depression and anxiety severity. These self-reports return scores indicative of momentary mental state. Self-reports are obtained intermittently from the participants.
Fear of Negative Evaluation Brief | 7-10 days
  Momentary self-reports of Fear of Negative Evaluation Brief will be administered in a tablet-based application. These self-reports return scores indicative of momentary mental state. Self-reports are obtained intermittently from the participants.

SECONDARY OUTCOMES:
Physiological measurements - heart rate variability (HRV) | 7-10 days
  Heart rate variability will be collected from each participant by using either commercial systems or the new wearable sensor.
Physiological measurements - skin conductance (SC) | 7-10 days
  Skin conductance will be collected from each participant by using either commercial systems or the new wearable sensor.
Physiological measurements - cortisol level | 7-10 days
  Cortisol level will be collected from each participant by using either commercial systems or the new wearable sensor.
Neural measurements | 7-10 days
  In epilepsy patients who already have intracranial EEG recordings for their standard clinical monitoring (unrelated to this study), we will also obtain iEEG activity measurements. EEG power will be the main focus of the analysis, but the raw signal will also be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shanechi, PhD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study and after publication, fully de-identified IPD may be made available for research purposes.
Time Frame: Any sharing will happen upon completion of the study and after publication.